CLINICAL TRIAL: NCT06873243
Title: Developing a Learning Health System to Address the Growing Burden of Noncommunicable Diseases in Thailand
Brief Title: Developing a Learning Health System for Primary Care in Thailand
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Royal Thai Ministry of Public Health (Unknown); London School of Hygiene and Tropical Medicine (Other); Chiang Mai University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0765; NIHR156161 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Diabetes; Kidney Disease; Primary Care; Primary Care Patients With Chronic Conditions; Quality Improvement
Keywords: Learning Health System; Quality Improvement; Hypertension; Diabetes; Kidney Disease; Primary Care; Non-Communicable Disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Kidney Diseases; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: We will conduct a three-phase open-label stratified cluster randomized controlled trial across two provinces in Thailand. Stratified randomisation will be used to allocate 16 primary care units from 419 total eligible primary care units to receive the intervention. We will generate four strata (the maximum number recommended for stratified cluster randomized trials of this size). Four primary care units in each stratum will be randomly selected to receive the intervention, and the rest will receive routine care (approximately 100 primary care units per stratum).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning Health System Intervention (Experimental): The intervention is the introduction of a Learning Health System approach to improve the management of hypertension, diabetes, and chronic kidney disease. The trial will encompass three of the four key components of complex intervention design: development of an intervention, assessment of feasibility of the intervention, and evaluation of the intervention.
  Primary care units randomized in the intervention will receive monthly data on their performance and patient outcome data from the CMU team. The data produced will be fed-back to practices via regular network-based peer discussions in a visually accessible format and facilitated by the clinical and community champions.
  Interventions: Behavioral: Learning Health System Approach
- Routine Care (No Intervention): This arm encompasses all primary care units not randomized to receive the intervention. Primary care units not randomized to the intervention will deliver routine care for hypertension, type 2 diabetes, and CKD. While we will collect monthly data on practice performance and key outcome metrics, they will not receive feedback or facilitation.

INTERVENTIONS:
Behavioral: Learning Health System Approach — Our intervention will be informed by the framework for designing LHSs developed by The Health Foundation and the updated framework for developing and evaluating complex evaluations commissioned by the UK Medical Research Council and National Institute for Health Research.The updated framework considers not only if an intervention is effective, but also whether the intervention is acceptable, implementable, cost-effective, scalable, and transferrable across contexts. The trial will encompass three of the four key components of complex intervention design: Development of an intervention Assessment of feasibility of the intervention, and Evaluation of the intervention. . We anticipate that a Plan Do Study Act (PDSA) cycle of quality improvement will be most suited to the Thai context as this approach is currently being promoted by the Thai Ministry of Public Health.
  Arms: Learning Health System Intervention

SUMMARY:
Research question: Can a Learning Health System (LHS) approach improve delivery of care and reduce inequalities in outcomes for people with hypertension and related non-communicable diseases (NCDs) compared to routine care in primary care settings in Thailand?

Background: NCDs account for 74% of all deaths in Thailand. Electronic health record data is used in Thailand to monitor how well whole regions deliver care, but is not directly available to healthcare teams in an actionable format which allows them to identify individuals in need of earlier, or more active management. LHS' are an effective framework for empowering healthcare teams to drive quality improvement (QI), reduce inequalities, and translate electronic health record data into actionable clinical insight.

Aims and objectives: We will conduct a stratified cluster randomized controlled trial to compare the LHS approach to routine care in two Thai provinces. We will randomize 16 primary care units to the intervention over three phases: targeting management of people with hypertension in phase 1, type 2 diabetes in phase 2 and chronic kidney disease (CKD) in phase 3. In each phase, we will: 1. Co-design a LHS with healthcare teams, policymakers, researchers and the public 2. Train healthcare and analytic teams to deliver the LHS and establish local champions to support it 3. Trial the LHS approach for 12 months 4. Compare performance between intervention and control practices and evaluate the benefits and costs of implementing the LHS 5. Identify provider and patient barriers and facilitators to inform long-term QI for NCDs

Methods: We will create four strata of primary care units according to practice size and case-mix. Within each stratum, we will randomize four practices to the intervention arm. In each of the three phases of the intervention, we will hold a series of stakeholder workshops to co-design quality improvement pathways, training materials, and computerised decision support tools (Aim 1); We will train multidisciplinary healthcare, analytic and research teams to implement the LHS and establish clinical and community champions to support it (Aim 2); We will trial the LHS for 12 months. Monthly data on key metrics will be used to monitor progress and iterate the LHS based on data analytics and shared learning across healthcare teams (Aim 3). We will conduct formal statistical comparisons between intervention and control arms, undertake health economic and mixed-methods realist evaluations to understand what works in promoting change and associated costs and benefits. (Aims 4 & 5).

Timeline: Trial setup (months 0-6), Hypertension (months 3-21), Diabetes (months 15-33), CKD (months 24-45), Evaluation (months 24-48)

Impact and dissemination: Results will be disseminated via publication in high-impact journals, conference presentations, stakeholder meetings, and the media. We will co-produce locally relevant educational materials and clinical guidelines. Impact will include the generation of longitudinal epidemiological data on management and outcomes of NCDs, including factors which facilitate continuous QI, and associated costs and benefits. The decision support tools, training resources, and economic evaluative frameworks will be made freely available by the Thai Ministry of Health and the regional WHO office. Capacity building will ensure the next generation of clinical, community, and research leaders promulgate this way of working across the region.

DETAILED DESCRIPTION:
Aims and objectives The overall aim of this study is to conduct a stratified cluster randomized controlled trial to determine whether a Learning Health System approach improves delivery of care and clinical outcomes for people with hypertension and related non-communicable diseases compared to routine care in primary care settings in Thailand. The trial will have three phases. In phase 1 we will trial an intervention for the management of people with hypertension. In phase 2 we will target the management of people with Type 2 Diabetes. In phase 3 we will target the management of people with CKD.

The key objectives for each phase of the intervention will be to:

1. Engage with healthcare providers, decision makers, researchers, and the public to co-design a LHS for the management of hypertension, diabetes, and CKD, and develop computerised data systems, decision support tools, and training materials in 16 randomly selected primary care units across two provinces in Thailand.
2. Train multidisciplinary healthcare teams, data scientists, and researchers in the design, delivery, analysis, and evaluation of a LHS and establish a cohort of clinical and community champions to support the intervention.
3. Pilot the delivery of a LHS for improving management and clinical outcomes of hypertension and related NCDs and generate robust new evidence around the acceptability and effectiveness of LHS approaches and delivery of clinical care.
4. Compare outcomes between intervention and control practices and conduct a health economic evaluation of the costs of implementing the LHS versus routine care.
5. Conduct a mixed-methods evaluations to identify provider and patient barriers and facilitators to implementing a LHS to inform subsequent approaches to embedding quality improvement for NCD care in Thai primary care settings and more widely across the region.

Our hypotheses are that:

1. Practices implementing the LHS approach will experience improved delivery of care and outcomes for people with hypertension, type 2 diabetes, and CKD vs. routine care
2. Training a multidisciplinary workforce and developing leadership capacity will embed continuous quality improvement approaches into routine clinical practice beyond the lifespan of this project

Research plan / methods Study Design: We will conduct a three-phase open-label stratified cluster randomized controlled trial across two provinces in Thailand. Stratified randomisation will be used to allocate 16 primary care units from 419 total eligible primary care units to receive the intervention (273 units in Chiang Mai and 146 units in Lampang). We will firstly stratify all primary care units in the study area according to patient population size (large vs. small practices) and patient case-mix (i.e. proportion of patients with any of hypertension, diabetes, and CKD), to ensure that primary care units within each stratum are balanced according to key characteristics. This will generate four strata (the maximum number recommended for stratified cluster randomized trials of this size29). Four primary care units in each stratum will be randomly selected to receive the intervention, and the rest will receive routine care (approximately 100 primary care units per stratum) Our intervention will be an open-label trial as those receiving the intervention will be aware of their allocation. We will register the trial with ClinicalTrials.gov and publish a trial protocol and statistical analysis plan prior to starting the study.

Phased approach of the intervention: The LHS intervention will have three distinct phases. In phase 1 we will design and implement a LHS for improving management of people with hypertension. In phase 2 we will design and implement a LHS for improving management of people with type 2 diabetes. In phase 3 we will design and implement a LHS for improving the management of people with CKD. The implementation of each phase will last 12 months.

Workstream 1: Co-designing the Learning Health System Intervention LHSs are complex and must be co-designed with local stakeholders. In addition to the project team, stakeholders will include: the healthcare teams (physicians, nurses, pharmacists, volunteer health workers); patients and members of the public; the Thai Ministry of Public Health (at national, provincial, and district level); the Thai World Health Organization; and the Thai Primary Care Support Office. Together the stakeholders will form a learning community who will drive the work of the LHS. The learning community will come together three times to co-design the LHS for each of the three phases of the intervention.

In collaboration with the stakeholder learning community, we will co-create computerised tools to support continuous monitoring, evidence generation, and quality improvement informed by electronic health record data. Tool development and data analysis will be led by the data science team at CMU. Tools will be tested and iterated upon by the learning community and healthcare teams throughout the life of the project.

In order to build capacity in embedding a culture of quality improvement into routine clinical care and data analytics, stakeholders will co-develop training modules to train healthcare teams on the design and implementation of LHSs.

Workstream 2: Training the multidisciplinary healthcare and research workforce and establishing clinical and community champions

Sourcing from each of the intervention practices, we will train a network of clinical and community champions who will support the intervention practices to deliver the LHS in the intervention practices. In partnership with the clinical and community champions, the team at CMU will deliver training to multidisciplinary healthcare and research teams in how to use quality improvement approaches for managing hypertension and related NCDs, use of computerised tools for routine monitoring, and translation of evidence into clinical action.

Workstream 3: Trialling implementation of the Learning Health System

Healthcare teams will implement the LHS approach agreed during the stakeholder consultation. They will be encouraged to meet regularly to discuss barriers and facilitators to implementing the LHS approach, to freely discuss problems they are experiencing, and to work collaboratively to diagnose and solve problems.

Healthcare teams will receive monthly data on their performance and patient outcome data from the CMU team. The data produced will be fed-back to practices via regular network-based peer discussions in a visually accessible format and facilitated by the clinical and community champions. Here, the practices will come together to review the data and share experiences of activities undertaken to improve care.

Primary care units not randomized to the LHS intervention will deliver routine care for hypertension, type 2 diabetes, and CKD. While we will collect monthly data on practice performance and key outcome metrics, they will not receive feedback or facilitation.

Workstream 4: Conducting quantitative comparisons between intervention and control primary care units and Health Economic Evaluation

All primary care units in the two participating Thai provinces will be included in the primary analysis according to their group assignment and regardless of their degree of participation in the study (intention-to-treat analysis). We will first conduct baseline comparisons of the intervention and control primary care units. While outcome data will be collected monthly, we will only conduct the formal evaluation for each phase of the intervention after the entire 12-month implementation period has elapsed. For phase 1, we will test the difference in the proportions of patients with hypertension meeting BP control targets between the intervention and control groups using a two-level generalized linear mixed-effects model which will account for the clustering of individuals within primary care units. We will repeat this approach for phase 2 (difference in the proportions of patients with type 2 diabetes meeting HbA1c control targets) and phase 3 (difference in the proportions of patients with CKD1-4 tested for albuminuria).

Health Economic Evaluation: We will develop an evaluation framework informed by Thai population data to support the evaluation of medium and long-term effects of the interventions implemented in the LHS. The project will make use of several unique large administrative databases including individual participant health data from Thai primary care and hospital systems. There will be three key patient populations of interest: people with hypertension, people with diabetes, and people with CKD. Therefore, we will develop an interactive Markov type decision-analytic model management of hypertension, diabetes and CKD using practice level factors, patient socio-demographic factors, clinical characteristics (e.g., systolic, and diastolic blood pressure, HbA1c, eGFR) and other risk factors (comorbidities). We will report reductions in disease risks, quality-adjusted life years gained and additional cost per quality-adjusted life year gained with interventions over medium term (5-10 years) and over lifetime.

Workstream 5: Conducting Realist Evaluation of the Learning Health System

We will undertake a realist evaluation of the programme alongside the trial to understand what works in promoting change, for whom, in what circumstances, how and why. The evaluation will include both quantitative and qualitative data collection and analyses to generate an overarching programme theory and identify the underlying causal mechanisms. We will start by generating an initial programme theory through an online interactive workshop drawing on learning and evidence gained from Workstream 1 and 2 activities. All research members and key stakeholders from the UK and Thailand will join the workshop. This initial programme theory will hypothesise how learning health systems in specific contexts (C), will trigger mechanisms (M) to generate outcomes (O).

We will collate the monthly quantitative data from the 16 intervention sites and all control sites within the same strata gathered by CMU throughout the intervention. Qualitative data collection will include gathering relevant documents for analysis and conducting focus groups. We will collate local documentation, such as board reports and minutes of meetings to understand the written outputs from QI activities. We will also collect qualitative data in a series of focus groups. We will undertake a document analysis of minutes from meetings and QI project reports. This process will lead to the development of an overall programme theory exploring if learning health systems work, in what circumstances, how and why.

ELIGIBILITY:
Inclusion Criteria:

* Any primary care unit in Lampang or Chiang Mai Province

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Hypertension | 12 months
  The proportion of adults with hypertension whose blood pressure meets target levels (<140/90 mmHg) at 12 months
Phase 2: Type 2 Diabetes | 12 months
  The proportion of adults with type 2 diabetes whose blood glucose meets target levels (<6.5%/48 mmol/mol) at 12 months
Phase 3: Chronic Kidney Disease | 12 months
  The proportion of adults with CKD stages 1-4 who are tested for albuminuria at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Mathur, PhD, Principal Investigator — Queen Mary University of London; Chaisiri Angkurawaranon, PhD, Principal Investigator — Chiang Mai University
Locations (1):
- Chiang Mai University, Chiang Mai, Chiang Mai District, Thailand

IPD SHARING:
Plan to Share IPD: No
The study is using routinely collected electronic health record data which is governed by the Thai Ministry of Health and not available for public release or re-use.